CLINICAL TRIAL: NCT04633863
Title: Pilot Study on Safety and Performance of an Artificial Tear Containing Arabinogalactan, Trehalose and Hyaluronic Acid in the Treatment of Dry Eye in Subjects With Inflammation of the Ocular Surface
Brief Title: Study on Safety and Performance of an Artificial Tear in Dry Eye Treatment in Subjects With Ocular Surface Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MD Italy (Industry)
Collaborators: Hippocrates Research (Other); Nubilaria Srl (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDI - 101
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDI - 101 (Experimental): Artificial tear containing arabinogalactan, trehalose and hyaluronic acid
  Interventions: Device: Artificial tear MDI - 101

INTERVENTIONS:
Device: Artificial tear MDI - 101 — Medical device CE marked - artificial tears containing arabinogalactan, trehalose and hyaluronic acid - 10 weeks treatment

SUMMARY:
This is post-market study to evaluate the safety and efficacy of MDI - 101 a novel tear substitute for the treatment of dry eye (DE) in subjects with evidence of inflammation of the ocular surface. In particular, this study intends to evaluate, in a cohort of 25 patients, the anti-inflammatory properties of the product under study over a period of 10 weeks

DETAILED DESCRIPTION:
DE is a common eye condition that affects 1 to 2 out of 10 persons in the world. Regardless of the underlying ethology, DE is associated with increased inflammation of conjunctiva, cornea and adnexa. As consequence of the recognized role of the inflammation in the etiopathogenesis of DE, direct and indirect anti-inflammatory treatments are currently the cornerstone for the management of DE, leading to the inhibition of the expression of inflammatory mediators on the ocular surface, therefore restoring the secretion of a healthy tear film and consequently reducing signs and symptoms of DE.

MDI - 101, the product under study containing arabinogalactan (AG), trehalose and hyaluronic acid (HA) ,is a medical device with European Conformity (CE) mark that, thanks to the muco-adhesive proprieties of AG enriches the natural mucous of the tear film providing enhanced lubrication and protection and anti-inflammatory properties, in combination with trehalose and HA. The aim of this study is to demonstrate that the reduced ocular discomfort and the improvement of the integrity of the ocular surface are due to the interruption of the "vicious cycle of inflammation".

This open-label study involves a cohort of 24 patients with clinical and instrumental signs of inflammation of the ocular surface and includes end-points of efficacy, safety and evaluation of inflammation markers. The study includes 6 visits over 10 weeks, 8 of which of active treatment. This study is conducted during the Covid-19 pandemic and for this reason, clinical assessments of all the 24 patients are carried out remotely, from patients' home, with the adoption of digital solutions that determine: reduction of 66% of physical contacts between investigator and patient, a total of 90% of efficacy and safety data collected remotely and a reduction of 100% of physical contacts between investigator and clinical monitor, keeping the study entirely within the Good Clinical Practice framework.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who gave their written consent for participation in the study and for personal data processing and willing to comply with all study procedures.
2. Males or females 30-75 years old.
3. Subjects who are familiar with the needs of the study in the use of mobile devices and internet.
4. Subjects who successfully completed the electronic registration for the clinical trial using their own study electronic Patient Reported Outcome (ePRO) profile and completed the OSDI questionnaire.
5. Subjects who had been diagnosed as having dry eye symptoms for at least 3 months, fulfilling all the following four criteria:

   i. OSDI score of >18 evaluated by the questionnaire of Ocular Surface Disease Index (OSDI); ii. Non-invasive breakup time (NIBUT) ≤10 seconds at least in one eye; iii. Levels of MMP-9 in tears ≥ 40 ng/ml as assessed by the Inflammatory assay at least in one eye; iv. Cornea surface scores ≥1 and <4, based on Efron grading system. -

Exclusion Criteria:

1. Contact lens wearers.
2. Subjects who did use any artificial tear for at least 7 days before baseline.
3. Severe corneal damage (cornea surface scores ≥4, based on Efron grading system) or cornea surface normal (scores <1 based on Efron grading system)
4. Corneal abrasions or other corneal abnormalities, blepharitis, meibomitis, lid abnormalities.
5. Conjunctivitis of infective or allergic origins, ongoing or resolved less than 4 weeks before baseline visit.
6. Subjects participating in another clinical study, on-going or completed less than 4 weeks before.
7. Subject using, or will use during the study, other artificial tear or other ophthalmic products including, but not limited, to: corticosteroids, antibiotics, vasoconstrictor agents.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy - Ocular Surface Disease Index (OSDI) | 1 week - 2 weeks - 4 weeks - 6 weeks - 8 weeks
  Change of OSDI score versus baseline at any study time-point. The main goal of the study is to gather information about the efficacy, assessed by OSDI (Ocular Surface Disease Index) questionnaire, of artificial tear containing AG, trehalose and HA (MDI - 101) used in the treatment of symptoms of DE of various aetiology, with evidence of inflammation of the ocular surface. The OSDI score ranges from 0 (better outcome) to 100 (worst outcome)

SECONDARY OUTCOMES:
Additional efficacy parameters: Matrix Metalloproteinase 9 (MMP-9) | 8 weeks
  Change of tear matrix metalloproteinase(MMP)-9 at T0 vs final assessment. The result of the MMP test could be NEGATIVE if the level of MMP-9 is < 40 ng/ml (better outcome) or POSITIVE if the level of MMP-9 is ≥ 40 ng/ml (worst outcome)
Additional Efficacy parameters: EFRON SCALE | 8 weeks
  Change of Efron Grading Scales at T0 vs final assessment. The Efron grading scale range from 0 (cornea surface normale) to 4 (severe corneal damage)
Additional Efficacy parameters: Corneal and Conjunctival Staining | 8 weeks
  Change of Corneal and Conjunctival Staining at T0 vs final assessment. The Staining scale ranges from 0 (better outcome) to 3 (worst outcome)
Additional Efficacy parameters: NIBUT | 8 weeks
  Change of NIBUT at T0 vs final assessment. The result of the Non-Invasive Break-Up Time (NIBUT) test could be >10 seconds (better outcome) or ≤10 seconds (worst outcome)
Additional Efficacy parameters: Osmolarity | 8 weeks
  Change of Osmolarity at T0 vs final assessment. The higher the tear film osmolarity, the greater the severity of the ocular surface damage.
Additional Efficacy parameters: Ocular Protection Index | 8 weeks
  Change of Ocular Protection Index (OPI) at T0 vs final assessment The principle of the test is that when BUT is shorter than the blink interval, the eyes are exposed to the risk of focal ocular surface damage.
Additional Efficacy parameters: meniscometry | 8 weeks
  Change of meniscometry at T0 vs final assessment. The lowest tear meniscus radius, the higher the severity of the ocular surface health
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 8 weeks
  Safety Adverse Event (AE) experienced with the artificial tear assessed by the patient, before the ocular examination or reported by the patient at any time during the study.
Incidence of change in the unaided and corrected visual acuity | 8 weeks
  Unaided and corrected visual acuity Snellen test will be performed to evaluate change in the unaided and corrected visual acuity at T0 vs final assessment.
Incidence of change in the Intraocular pressure | 8 weeks
  Change of Intraocular pressure at T0 vs final assessment.
Evaluation of the Tolerability Signs and symptoms of discomfort | 8 weeks
  Treatment adherence assessed by the patient at any study time-point (number of instillations in the past 24 hours).
Treatment adherence (24 hours) | 8 weeks
  Treatment adherence assessed by the patient at any study time-point (number of instillations in the past 24 hours)
Treatment adherence (total days) | 8 weeks
  Treatment adherence assessed by the patient at any study time-point (number of days of product usage).

CONTACTS AND LOCATIONS:
Overall Officials: Ophthalmology unit, Principal Investigator — Lucca
Locations (1):
- Ophthalmology unit, Lucca, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Battelli MG, Bolognesi A, Polito L. Pathophysiology of circulating xanthine oxidoreductase: new emerging roles for a multi-tasking enzyme. Biochim Biophys Acta. 2014 Sep;1842(9):1502-17. doi: 10.1016/j.bbadis.2014.05.022. Epub 2014 May 29. PMID 24882753
- [Result] Baudouin C. [A new approach for better comprehension of diseases of the ocular surface]. J Fr Ophtalmol. 2007 Mar;30(3):239-46. doi: 10.1016/s0181-5512(07)89584-2. French. PMID 17417148
- [Result] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Result] Burgalassi S, Nicosia N, Monti D, Falcone G, Boldrini E, Chetoni P. Larch arabinogalactan for dry eye protection and treatment of corneal lesions: investigations in rabbits. J Ocul Pharmacol Ther. 2007 Dec;23(6):541-50. doi: 10.1089/jop.2007.0048. PMID 18001233
- [Result] Cejka C, Kubinova S, Cejkova J. Trehalose in ophthalmology. Histol Histopathol. 2019 Jun;34(6):611-618. doi: 10.14670/HH-18-082. Epub 2019 Jan 9. PMID 30623968
- [Result] Choy CK, Cho P, Boost MV. Cytotoxicity of rigid gas-permeable lens care solutions. Clin Exp Optom. 2013 Sep;96(5):467-71. doi: 10.1111/cxo.12039. Epub 2013 May 3. PMID 23638722
- [Result] Efron N, Morgan PB, Jagpal R. Validation of computer morphs for grading contact lens complications. Ophthalmic Physiol Opt. 2002 Jul;22(4):341-9. doi: 10.1046/j.1475-1313.2002.00049.x. PMID 12162486
- [Result] Kelly GS. Larch arabinogalactan: clinical relevance of a novel immune-enhancing polysaccharide. Altern Med Rev. 1999 Apr;4(2):96-103. PMID 10231609
- [Result] Hessen M, Akpek EK. Dry eye: an inflammatory ocular disease. J Ophthalmic Vis Res. 2014 Apr;9(2):240-50. PMID 25279127
- [Result] Holden BA, Reddy MK, Sankaridurg PR, Buddi R, Sharma S, Willcox MD, Sweeney DF, Rao GN. Contact lens-induced peripheral ulcers with extended wear of disposable hydrogel lenses: histopathologic observations on the nature and type of corneal infiltrate. Cornea. 1999 Sep;18(5):538-43. PMID 10487426
- [Result] Jain NK, Roy I. Effect of trehalose on protein structure. Protein Sci. 2009 Jan;18(1):24-36. doi: 10.1002/pro.3. PMID 19177348
- [Result] Li W, Sun X, Wang Z, Zhang Y. A survey of contact lens-related complications in a tertiary hospital in China. Cont Lens Anterior Eye. 2018 Apr;41(2):201-204. doi: 10.1016/j.clae.2017.10.007. Epub 2017 Oct 21. PMID 29033270
- [Result] Pahuja P, Arora S, Pawar P. Ocular drug delivery system: a reference to natural polymers. Expert Opin Drug Deliv. 2012 Jul;9(7):837-61. doi: 10.1517/17425247.2012.690733. Epub 2012 Jun 16. PMID 22703523
- [Result] Shi YH, Zhou LT, Zhang CX, Li YZ, Zhang JZ, Zhou HM, Li YG, Liu T, Zhang LL, Sun LN, Chen Z. Effects of carbomer eye drops in combination with orthokeratology lens in treating adolescent myopia. J Biol Regul Homeost Agents. 2016 Oct-Dec;30(4):1029-1033. PMID 28078849
- [Result] Silvani L, Bedei A, De Grazia G, Remiddi S. Arabinogalactan and hyaluronic acid in ophthalmic solution: Experimental effect on xanthine oxidoreductase complex as key player in ocular inflammation (in vitro study). Exp Eye Res. 2020 Jul;196:108058. doi: 10.1016/j.exer.2020.108058. Epub 2020 May 4. PMID 32380019
- [Result] Stuart JC, Linn JG. Dilute sodium hyaluronate (Healon) in the treatment of ocular surface disorders. Ann Ophthalmol. 1985 Mar;17(3):190-2. PMID 3873200
- [Result] Sullivan DA, Rocha EM, Aragona P, Clayton JA, Ding J, Golebiowski B, Hampel U, McDermott AM, Schaumberg DA, Srinivasan S, Versura P, Willcox MDP. TFOS DEWS II Sex, Gender, and Hormones Report. Ocul Surf. 2017 Jul;15(3):284-333. doi: 10.1016/j.jtos.2017.04.001. Epub 2017 Jul 20. PMID 28736336
- [Result] Yokoi N, Komuro A. Non-invasive methods of assessing the tear film. Exp Eye Res. 2004 Mar;78(3):399-407. doi: 10.1016/j.exer.2003.09.020. PMID 15106919